CLINICAL TRIAL: NCT02950831
Title: Objective Assessment of Activity and Sleep Quality In Burst Spinal Cord Stimulation
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: AZ Sint-Augustinus, Wilrijk (Unknown); AZ Middelheim, Antwerpen (Unknown); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJM-CIP-10133
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; BurstDR; spinal cord stimulation; Accelerometry
MeSH Terms: conditions — Chronic Pain | interventions — Accelerometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activity and sleep quality recording (Experimental): Patients will receive a wrist worn accelerometer and accelerometry will be used to monitor physical activity and sleep quality during standard BurstDR Spinal Cord Stimulation clinical treatment
  Interventions: Other: Accelerometry

INTERVENTIONS:
Other: Accelerometry — Record of activity levels using a wrist worn accelerometer
  Other Names: wrist worn accelerometers

SUMMARY:
The purpose of this study is to assess feasibility of using wearable sensors to capture objective assessments of patient's activity and sleep quality during the spinal cord stimulation (SCS) treatment continuum.

DETAILED DESCRIPTION:
Eligible patients will undergo standard clinical care using BurstDR SCS and will be asked to wear a wrist worn accelerometer for a baseline period, during SCS trial and for 3 months after activation of the SCS stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent to participate in the study;
* Subject is 18 years of age or older;
* Subject has failed to respond to at least 6 months of conventional treatment including pharmacological treatment, physical therapy, epidural injections and/or radiofrequency therapy;
* Subjects with the diagnosis of failed back surgery syndrome or chronic intractable trunk and/or lower limb pain and are eligible for a SCS trial;
* Subjects have an average trunk pain VAS score of at least 6.0 out of 10.0, and/or lower limb pain VAS score of at least 6.0 out of 10.0;
* Subject is on stable pain medications, as determined by the Investigator, for at least 28 days prior to enrolling in this study, and is willing to stay on those medications with no dose adjustments until activation of the permanently implanted SCS device;
* Subject's medical record has been evaluated by the Investigator to ensure that the subject is a good candidate for a neurostimulation system;
* Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all office visits;
* Subject agrees to wear the wearable sensor for the duration of the study;
* Female candidates of child-bearing potential agree to commit to the use of an effective method of contraception (including but not limited to sterilization, barrier devices, oral contraceptives, intrauterine devices (IUDs), condoms, rhythm method, or abstinence) for the duration of the study

Exclusion Criteria:

* Subject is currently participating in a clinical investigation that includes an active treatment arm;
* Subject has been implanted with or participated in a trial period for a neurostimulation system;
* Non- ambulatory subjects who are not expected to become ambulatory after receiving neurostimulation;
* Subject diagnosed with fibromyalgia or chronic fatigue;
* Subject has an infusion pump;
* Subject has evidence of an active disruptive psychological or psychiatric disorder as determined as per standard of care;
* Subject has a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease or uncontrolled diabetes mellitus;
* Subject has a current diagnosis of a progressive neurological disease as determined by the Investigator;
* Subject is immunocompromised;
* Subjects with concurrent clinically significant or disabling chronic pain problem that requires additional treatment;
* Subject has an existing medical condition that is likely to require repetitive MRI evaluation in the future (i.e. epilepsy, stroke, multiple sclerosis, acoustic neuroma, tumor);
* Subject has history of cancer requiring active treatment in the last 12 months;
* Subject has an existing medical condition that is likely to require the use of diathermy in the future;
* Subject has documented history of allergic response to titanium or silicone;
* Subject has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the 6 months prior to baseline data collection;
* Female candidates of child bearing potential that are pregnant (confirmed by positive urine/blood pregnancy test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lalit Venkatesan, Ph.D., Study Director — Abbott Medical Devices
Locations (3):
- Belgium (2):
  - AZ Sint-Augustinus, Wilrijk, Antwerp
  - AZ Middelheim, Antwerp, Flanders
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activity and Sleep Quality Recording
Started | 27
Complete Trial | 26
Permanent Implant | 20
4 Week Follow up | 20
8 Weeks Follow up | 19
Completed | 18
Not Completed | 9
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — stimulation trail failure | 5

BASELINE CHARACTERISTICS:
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 27
Region of Enrollment [Number; unit: participants]
  Netherlands | 22
  Belgium | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Activity Levels
Description: Recording performed with wrist worn accelerometer. Medium to Vigorous Physical Activity (MVPA) were calculated based on accelerometry data. MVPA value represents the hours of medium to vigorous physical activity in a day.
Time Frame: between baseline and the end of spinal cord stimulation trial period (average of 1 month)
Population: Average change in MVPA (h/day) from baseline value is reported. Activity recording files were not available for 2 patients.
Measure: Mean (Standard Deviation); unit: change in MVPA h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 24
change in MVPA h/day from baseline value | -0.17 (0.22)

2. Primary Outcome: Change in Sleep Quality
Description: Recording performed with wrist worn accelerometer. Sleep duration was calculated based on accelerometry data.
Time Frame: between baseline and the end of spinal cord stimulation trial period (average of 1 month)
Population: Change in average sleep duration from baseline value is reported. Activity recording files were not available for 2 patients.
Measure: Mean (Standard Deviation); unit: Change h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 24
Change h/day from baseline value | -0.05 (1.05)

3. Secondary Outcome: Change in Visual Analog Scale (VAS) for Pain
Description: Subjective evaluation of pain levels used in clinical practice as standard. Minimum value is 0 (no pain), maximum value is 10 (maximum pain imaginable)
Time Frame: between baseline and the end of spinal cord stimulation trial period (average of 1 month)
Population: Percentage change in average VAS value from baseline is reported (pain relief) Data was not available for 1 subject
Measure: Mean (Standard Error); unit: Percentage reduction from baseline score
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 25
Percentage reduction from baseline score | -57.73 (31.4)

4. Secondary Outcome: Change in Visual Analog Scale (VAS) for Pain
Description: as for outcome 3
Time Frame: between baseline and 1 month post permanent spinal cord stimulator activation followup
Population: Percentage reduction in average VAS value from baseline is reported (pain relief)
Measure: Mean (Standard Error); unit: Percentage change from baseline score
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 20
Percentage change from baseline score | -49.04 (47.49)

5. Secondary Outcome: Change in Visual Analog Scale (VAS) for Pain
Description: as for outcome 3
Time Frame: between baseline and 2 month post permanent spinal cord stimulator activation followup
Population: Percentage change in average VAS value from baseline is reported (pain relief)
Measure: Mean (Standard Deviation); unit: Percentage reduction from baseline score
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 19
Percentage reduction from baseline score | -53.55 (43.81)

6. Secondary Outcome: Change in Visual Analog Scale (VAS) for Pain
Description: as for outcome 3
Time Frame: between baseline and 3 month post permanent spinal cord stimulator activation followup
Population: Percentage change in average VAS value from baseline is reported (pain relief)
Measure: Mean (Standard Deviation); unit: Percentage change from baseline score
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 18
Percentage change from baseline score | 52.04 (44.95)

7. Secondary Outcome: Change in European Quality of Life 5 Dimensions (EQ-5D)
Description: Questionnaire pertaining to quality of life. Minimum Value 0, maximum value 1 with higher numbers representing higher quality of life.
Time Frame: between baseline and the end of spinal cord stimulation trial period (average of 1 month)
Population: Change in average EQ-5D scores from baseline is reported
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 26
change in score on a scale | 0.23 (0.12)

8. Secondary Outcome: Change in European Quality of Life 5 Dimensions (EQ-5D)
Description: as for outcome 7
Time Frame: between baseline and 1 month post permanent spinal cord stimulator activation followup
Population: Change in average EQ-5D scores from baseline is reported
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 20
change in score on a scale | 0.19 (0.17)

9. Secondary Outcome: Change in European Quality of Life 5 Dimensions (EQ-5D)
Description: as for outcome 7
Time Frame: between baseline and 2 month post permanent spinal cord stimulator activation followup
Population: Change in average EQ-5D scores from baseline is reported
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 19
change in score on a scale | 0.23 (0.14)

10. Secondary Outcome: Change in European Quality of Life 5 Dimensions (EQ-5D)
Description: as for outcome 7
Time Frame: between baseline and 3 month post permanent spinal cord stimulator activation followup
Population: Change in average EQ-5D scores from baseline is reported
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 18
change in score on a scale | 0.18 (0.19)

11. Secondary Outcome: Change in Oswestry Disability Index (ODI)
Description: Questionnaire pertaining to disability levels. Minimum value 0, maximum value 100 with higher values representing higher levels of disability.
Time Frame: between baseline and the end of spinal cord stimulation trial period (average of 1 month)
Population: Percentage change in average ODI value from baseline is reported. One patient did not complete the ODI form correctly.
Measure: Mean (Standard Error); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 25
change in score on a scale | -18.6 (15.8)

12. Secondary Outcome: Change in Oswestry Disability Index (ODI)
Description: as for outcome 11
Time Frame: between baseline and 1 month post permanent spinal cord stimulator activation followup
Population: Change in average ODI value from baseline is reported.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 20
change in score on a scale | -17.4 (14.6)

13. Secondary Outcome: Change in Oswestry Disability Index (ODI)
Description: as for outcome 11
Time Frame: between baseline and 2 month post permanent spinal cord stimulator activation followup
Population: Change in average ODI value from baseline is reported.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 19
change in score on a scale | -18.8 (14.0)

14. Secondary Outcome: Change in Oswestry Disability Index (ODI)
Description: as for outcome 11
Time Frame: between baseline and 3 month post permanent spinal cord stimulator activation followup
Population: Change in average ODI value from baseline is reported.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 18
change in score on a scale | -19.1 (13.6)

15. Secondary Outcome: Change in Activity Levels
Description: Recording performed with wrist worn accelerometer. Medium to Vigorous Physical Activity (MVPA) were calculated based on accelerometry data. MVPA value represents the hours of medium to vigorous physical activity in a day.
  Average percent change in MVPA from baseline value is reported.
Time Frame: between baseline and 1 month post permanent spinal cord stimulator activation followup
Population: Average change in MVPA (h/day) from baseline value is reported. Activity recording files were not available for 1 patient
Measure: Mean (Standard Deviation); unit: change in MVPA h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 19
change in MVPA h/day from baseline value | -0.01 (0.09)

16. Secondary Outcome: Change in Sleep Quality
Description: Recording performed with wrist worn accelerometer. Sleep duration was calculated based on accelerometry data.
Time Frame: between baseline and 1 month post permanent spinal cord stimulator activation followup
Population: Change in average sleep duration from baseline value is reported. Activity recording files were not available for 1 patient
Measure: Mean (Standard Deviation); unit: Change h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 19
Change h/day from baseline value | 0.1 (0.82)

17. Secondary Outcome: Change in Activity Levels
Description: as for outcome 15
Time Frame: between baseline and 2 month post permanent spinal cord stimulator activation followup
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: change in MVPA h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 18
change in MVPA h/day from baseline value | 0.03 (0.08)

18. Secondary Outcome: Change in Sleep Quality
Description: Recording performed with wrist worn accelerometer. Sleep duration was calculated based on accelerometry data.
Time Frame: between baseline and 2 month post permanent spinal cord stimulator activation followup
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Change h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 18
Change h/day from baseline value | -0.06 (0.81)

19. Secondary Outcome: Change in Activity Levels
Description: as for outcome 15
Time Frame: between baseline and 3 month post permanent spinal cord stimulator activation followup
Population: Average change in MVPA (h/day) from baseline value is reported. Activity files were not available for 5 patients
Measure: Mean (Standard Deviation); unit: change in MVPA h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 13
change in MVPA h/day from baseline value | 0.02 (0.08)

20. Secondary Outcome: Change in Sleep Quality
Description: Recording performed with wrist worn accelerometer. Sleep duration was calculated based on accelerometry data.
Time Frame: between baseline and 3 month post permanent spinal cord stimulator activation followup
Population: Percent change in average sleep duration from baseline value is reported. Activity files were not available for 5 patients
Measure: Mean (Standard Deviation); unit: Change h/day from baseline value
Arm/Group | Activity and Sleep Quality Recording
Number analyzed (Participants) | 13
Change h/day from baseline value | 0 (0.61)

ADVERSE EVENTS:
Time Frame: From baseline to 3rd month follow up for an average duration of 4.6 months (including trial and wait time between trial and permanent implant)
Arm/Group | Activity and Sleep Quality Recording
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 3/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activity and Sleep Quality Recording (N=27)
Increased pain/inadequate pain relief that required device reprogramming (Nervous system disorders) | 2 (4)
IPG pocket pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT02950831/Prot_SAP_000.pdf